CLINICAL TRIAL: NCT01429103
Title: Hormones and Cognition in the Menopausal Transition
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Miriam Weber, Assistant Professor, University of Rochester
Other Study IDs: Weber K23; 1K23AG034256 (NIH)
Record Dates: First submitted 2011-09-01; First posted 2011-09-05 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Age-associated Memory Impairment; Alteration of Cognitive Function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Subjects will have 20 mL of blood drawn by venipuncture by a trained nurse
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Early Perimenopause: Early perimenopause is defined as the presence of irregular periods (cycle length differs by 7 days from usual).
- Late Perimenopause: Late perimenopause is defined as at least 2 skipped periods over the past 12 months (cycle double usual length) and one period of amenorrhea (over 60 days without a period), with at least one menstrual cycle over the past 12 months.

SUMMARY:
The purpose of this study is to determine if the menopausal transition is associated with subjective and objective cognitive declines that ameliorate in menopause. The investigators hypothesize that perimenopause is associated with both subjective memory complaints and objective declines in attentionally mediated cognitive tasks. The investigators also hypothesize that this is time-limited. The investigators predict that as women transition from early perimenopause to late perimenopause their performance on attentionally mediated and verbal memory tasks will decline, and that as they transition from late perimenopause to menopause, their performance will improve.

DETAILED DESCRIPTION:
Two groups of women will be recruited, those in early perimenopause and those in mid to late perimenopause. Tests of attention, working memory, mental flexibility, processing speed, and retentive memory will be administered to each subject at 6 month intervals for 5 years. Additionally, women will be asked to fill out questionnaires about their mood, memory functioning, health, and quality of life. The investigators will also calculate each subject's Body Mass Index (BMI) and waist circumference at each visit. Finally, serum levels of reproductive hormones will be taken. Measures of interest will be the percentage of women in each group with absolute and relative cognitive deficits, change over time in performance on neuropsychological tests and scores on depression and anxiety scales, and correlations between cognitive function, mood and hormone level.

ELIGIBILITY:
Inclusion Criteria:

Menopausal status will be based on self-report of menstrual cycles over the past 12 months. Early perimenopause is defined as the presence of irregular periods (cycle length differs by 7 days from usual). Late perimenopause is defined as at least 2 skipped periods over the past 12 months (cycle double usual length) and one period of amenorrhea (over 60 days without a period), with at least one menstrual cycle over the past 12 months, according to the Stages of Reproductive Aging Workshop criteria.

Exclusion Criteria:

- history of neurological disease known to affect cognitive function (i.e., stroke, MS, etc) and major psychiatric illness. The investigators will exclude women who are currently pregnant or breast-feeding, have undergone surgical menopause, or who have used exogenous hormone preparations affecting ovarian or pituitary function in the past 3 months. The investigators will also exclude women who have had hysterectomies, but intact ovaries, or oophorectomies. Women who choose to initiate HRT at some point during the study will continue to be followed, but their data obtained after HRT is initiated will be analyzed separately.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women between the ages of 40 and 60.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2011-05; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Weber, PhD, Principal Investigator — Department of Neurology, University of Rochester
Locations (1):
- University of Rochester Clinical Research Center, Rochester, New York, United States